CLINICAL TRIAL: NCT03787914
Title: Community Outreach Mobile Teams Impact on Tuberculosis Treatment Outcome in Jeddah Region: A Randomized Controlled Trial
Brief Title: Effect of Community Mobile Outreach Approach Compared to Facility Based Directly Observed Treatment Short Course on Treatment Outcome Among Tuberculosis Patients in Jeddah: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Hassan Bin Usman, Public Health Specialist, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-02-J-002-00877
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: The investigators conducted a two-arm, parallel design[1:1], single blind randomized control trial in 200 newly diagnosed TB patients
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Intervention arm patients were served by outreach mobile teams for oral anti-TB treatment under DOTS at the place of their convenience by health care professionals
  Interventions: Procedure: Mobile Outreach Approach
- Control arm (Active Comparator): Control arm patients were given the traditional facility based DOTS treatment. Control arm was not served by the outreach mobile teams.
  Interventions: Procedure: Mobile Outreach Approach

INTERVENTIONS:
Procedure: Mobile Outreach Approach — TB patients in intervention arm were served by outreach mobile teams for DOTS (i.e. administration of anti-TB medicines orally at the place and time of their choice and convenience under mobile teams direct supervision

SUMMARY:
To compare the effectiveness of the community mobile outreach approach in improving treatment outcomes (success rate) among tuberculosis patients with those being treated with facility based directly observed treatment short course (DOTS) in Jeddah region.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed TB cases

Exclusion Criteria:

* Visitors having TB especially pilgrims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Treatment Success rate | 6 to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah AlSahafi, MBBS, SBFM, Study Director — Director of Public Health
Locations (1):
- Ministry of Health, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Sahafi A, Al-Sayali MM, Mandoura N, Shah HBU, Al Sharif K, Almohammadi EL, Abdul-Rashid OA, Assiri M, Buksh MF, Alali MM, Al-Garni A, Al-Garni F, Al-Zahrani A, Khalawi A, Alawi M, Moawwad AL, Almalki AIA, Al-Osaimi MM. Treatment outcomes among tuberculosis patients in Jeddah, Saudi Arabia: Results of a community mobile outreach directly observed Treatment, Short-course (DOTS) project, compared to a standard facility-based DOTS: A randomized controlled trial. J Clin Tuberc Other Mycobact Dis. 2020 Dec 31;22:100210. doi: 10.1016/j.jctube.2020.100210. eCollection 2021 Feb. PMID 33490640